CLINICAL TRIAL: NCT01056354
Title: An International Observational Study to Characterize Adults With Influenza or Other Targeted Respiratory Viruses
Brief Title: Respiratory Virus Outpatient Study (FLU 002 Plus)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0603M83587 FLU 002; HHSN261200800001E ; 29XS214 (Other Grant/Funding Number: Science Applications International Corporation (SAIC))
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Influenza and Other Novel Respiratory Viruses
Keywords: Influenza; respiratory virus; pandemic; swine flu; infection; MERS-CoV; SARS-CoV
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections; Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Upper respiratory tract specimen
  Serum and plasma
  For participants with a confirmed targeted non-influenza respiratory virus, attempts will be made to obtain a sample of the local specimen used to confirm diagnosis.
  Whole blood for human genomics (only at FLU 002 Plus sites opting to also participate in INSIGHT Genomics and participant has signed an additional consent)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Influenza: Influenza A and subtypes such as H3N2 and 2009 H1N1 or influenza B
- Novel respiratory virus-1: MERS-CoV (Middle Eastern Respiratory Syndrome Coronavirus)
- Novel respiratory virus-2: SARS-CoV (Severe Acute Respiratory Syndrome Coronavirus)

SUMMARY:
Following the sudden and unexpected emergence of influenza A(H1N1)pdm09 (2009 H1N1) virus, this observational study was initiated to describe participants seeking medical care in geographically diverse locations with 2009 H1N1 infection and their clinical course over a 14-day period following enrollment. In 2011, as surveillance indicated that 2009 H1N1 virus was co-circulating with other seasonal influenza A and B viruses worldwide, the protocol was expanded to include other influenza A subtypes and influenza B viruses. This version of the protocol further broadens the scope of this observational study. With the recognition that novel respiratory viruses other than novel influenza A viruses, e.g., Middle East Respiratory Syndrome Coronavirus (MERS-CoV), could become prevalent and of major public health importance, the objectives of this protocol have been expanded

DETAILED DESCRIPTION:
The purpose of this observational study is to describe participants in geographically diverse locations with influenza virus infection and other viral respiratory diseases of public health importance and their clinical course over a 14-day period following enrollment.

Specific objectives related to influenza virus infection are to estimate the percentage of participants who go on to develop severe disease or complications that require hospitalization; to obtain information on risk factors for disease severity; and to establish a central repository of specimens for use in virus characterization, including subtyping, antigenic and genetic analyses, identification of signature mutations associated with antiviral drug resistance, mutational evolution, and additional reassortment.

Specific objectives related to novel non-influenza respiratory viruses of potential major public health importance are to characterize initial cases and their outcomes in order to develop more specific protocols that could inform the prevention and treatment of these new infections

Sample size is open-ended for this observational study. Based on experience to date, it is estimated that 75 sites will participate and will enroll approximately 1,700 patients with influenza each year, about one-half in the Northern Hemisphere and one-half in the Southern Hemisphere. Sites in diverse geographic locations on several continents will participate.

Study Plan:

* Participants who meet the eligibility criteria will be enrolled at participating clinical sites.
* At enrollment, consent is signed and information (demographics, medical history (including prior influenza and pneumococcal vaccination), medications (including antivirals) and treatments prescribed will be recorded. A blood sample for serum and plasma will be obtained at enrollment, as well as an upper respiratory tract specimen. The respiratory specimen will be sent for central reverse transcriptase polymerase chain reaction (RT-PCR) testing for influenza.
* Status will be re-assessed at approximately 14 days after enrollment and another blood sample for serum and plasma will be obtained. For participants with a confirmed novel respiratory virus of public health importance, attempts will be made to obtain a sample of the local specimen used to diagnose the infection.

In February 2012, the FLU 004 Genomics protocol v 1.0 was released to the field.

In August 2013 v 2.0 of the protocol was released as INSIGHT Genomics. The protocol was expanded beyond the FLU 002 and FLU 003 studies to include all qualifying INSIGHT studies (list posted on the INSIGHT website, www.insight-trials.org. The purpose of this substudy is to obtain a whole blood sample from which DNA will be extracted to study polymorphisms in immune response genes and other genetic variants that may be associated with an increased risk of disease progression among individuals with infectious diseases of public health importance who are enrolled in qualifying INSIGHT studies.

Participating FLU 002 Plus sites are given the option to also participate in INSIGHT Genomics, which requires a separate protocol registration. Participants, once consented to FLU 002 Plus, will be offered the option to also consent to INSIGHT Genomics, which includes a single whole blood sample collection. Participation in FLU 002 Plus will not be compromised if a participant opts not to participate in INSIGHT Genomics.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age
* Have a signed informed consent by participant
* Have a fever (37.8 degrees C (100 degrees F) or higher on examination or patient-reported fever (37.8 degrees C (100 degrees F) or higher, or feverishness (felt febrile but did not take temperature) in the past 24 hours.
* Have a cough and/or sore throat
* Have suspected influenza or a suspected targeted non-influenza viral respiratory infection

Exclusion Criteria:

- Current imprisonment, or compulsory detention (involuntary incarceration) for treatment of a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who seek medical care and are suspected of having influenza or a targeted novel respiratory virus* of major public health concern will be enrolled at numerous participating clinical sites on several continents.
  *The current list of other targeted novel respiratory viruses includes MERS-CoV and SARS-CoV.
Sampling Method: Probability Sample
Enrollment: 11719 (Actual)
Dates: Start 2009-08; Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Death or Hospitalization | 14-day period following enrollment
  Death or hospitalization within 14 days of enrollment or the development of one severe complication.

SECONDARY OUTCOMES:
Days of work/school lost, duration of symptoms, use of antivirals | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: James Neaton, Professor, Principal Investigator — University of Minnesota - Dept Biostatistics
Locations (68):
- United States (17):
  - UCSD Antiviral Research Center, San Diego, California
  - Denver Public Health, Denver, Colorado
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Infectious Diseases Associates NW FL, PA, Pensacola, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Newland Immunology Center of Excellence (NICE), Southfield, Michigan
  - New Jersey Medical School Adult Clinical Research Center, Newark, New Jersey
  - Cornell CRS, New York, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - UNC AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Tennessee College of Medicine, Chattanooga, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston AIDS Research Team, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (12):
  - Hospital Nacional Profesor Alejandro Posadas, El Palomar, Buenos Aires
  - Hospital Interzonal General de Agudos Dr. Diego Paroissien, La Matanza, Buenos Aires
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Hospital Profesor Bernardo Houssay, Vicente López, Buenos Aires
  - CAICI (Instituto Centralizado de Assistencia e Investigacion Clinica Integral), Rosario, Santa Fe Province
  - Sanatorio Britanico, Rosario, Santa Fe Province
  - CEMIC, Buenos Aires
  - FUNCEI, Buenos Aires
  - Hospital General de Agudos JM Ramos Mejia, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital Rawson, Córdoba
- Australia (5):
  - Interchange General Practice, Canberra, Australian Capital Territory
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Northside Clinic, Fitzroy North, Victoria
  - Prahran Market Clinic, Melbourne, Victoria
- Belgium (2):
  - Centre Hospitalier Universitaire St. Pierre (C.H.U. St. Pierre), Brussels
  - Practimed Medisch Centrum Tessenderlo, Tessenderlo
- Chile (3):
  - Clinica Alemana, Santiago
  - Fundacion Arriaran, Santiago
  - Pontificia Universidad Catolica de Chile, Santiago
- Denmark (4):
  - Arhus Universitetshospital, Skejby, Aarhus
  - CHIP, Copenhagen
  - Rigshospitalet, Infektionsmedicinsk ambulatorium 8622, Copenhagen
  - University Clinic of General Practice, Copenhagen
- West Tallinn Central Hospital Infectious Diseases, Tallinn, Estonia
- Germany (4):
  - Medizinische Universitatsklinik - Bonn, Immunologische Ambulanz CRS, Bonn
  - Klinik I fur Innere Medizin der Universitat zu Koln, Studienburo fur Infektiologie u. HIV, Cologne
  - Johann Wolfgang Goethe - University Hospital, Infektionsambulanz CRS, Frankfurt
  - Ifi - Studien und Projekte GmbH, Hamburg
- Greece (4):
  - 1st Dept of Critical Care Medicine and Pulmonary Services, Evangelismos Hospital, Athens
  - 1st Respiratory Medicine Dept, Athens Hosp for Diseases of the Chest "Sotiria Hospital", Athens
  - Evangelismos General Hospital, Athens
  - Hippokration University General Hospital of Athens, Athens
- National Hospital Organization Nagoya Medical Center, Nagoya, Japan
- Peru (4):
  - Hospital Nacional Arzobispo Loayza, Lima
  - Asociacion Civil IMPACTA Salud y Educacion, Lima
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Poland (2):
  - Wojewodzki Szpital Zakazny, Warsaw
  - EMC Instytut Medyczny SA, Wroclaw
- Spain (2):
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz
- Thailand (3):
  - Chulalongkorn University Hospital, Bangkok
  - Khon Kaen University, Srinagarind Hospital, Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi
- United Kingdom (4):
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Churchill Hospital, Headington, Oxford
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire
  - St James's University Hospital, Leeds, West Yorkshire

REFERENCES:
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] World Health Organization (WHO), www.who.int/, accessed 26 August 2013
- [Background] Guery B, Poissy J, el Mansouf L, Sejourne C, Ettahar N, Lemaire X, Vuotto F, Goffard A, Behillil S, Enouf V, Caro V, Mailles A, Che D, Manuguerra JC, Mathieu D, Fontanet A, van der Werf S; MERS-CoV study group. Clinical features and viral diagnosis of two cases of infection with Middle East Respiratory Syndrome coronavirus: a report of nosocomial transmission. Lancet. 2013 Jun 29;381(9885):2265-72. doi: 10.1016/S0140-6736(13)60982-4. Epub 2013 May 30. PMID 23727167
- [Background] Drosten C, Seilmaier M, Corman VM, Hartmann W, Scheible G, Sack S, Guggemos W, Kallies R, Muth D, Junglen S, Muller MA, Haas W, Guberina H, Rohnisch T, Schmid-Wendtner M, Aldabbagh S, Dittmer U, Gold H, Graf P, Bonin F, Rambaut A, Wendtner CM. Clinical features and virological analysis of a case of Middle East respiratory syndrome coronavirus infection. Lancet Infect Dis. 2013 Sep;13(9):745-51. doi: 10.1016/S1473-3099(13)70154-3. Epub 2013 Jun 17. PMID 23782859
- [Background] World Health Organization (WHO), Severe Acute Respiratory Syndrome (SARS), www.who.int/csr/sars/, accessed 26 August 2013
- [Derived] Simonsen L, Higgs E, Taylor RJ, Wentworth D, Cozzi-Lepri A, Pett S, Dwyer DE, Davey R, Lynfield R, Losso M, Morales K, Glesby MJ, Weckx J, Carey D, Lane C, Lundgren J; INSIGHT FLU002 and FLU003 Study Groups. Using Clinical Research Networks to Assess Severity of an Emerging Influenza Pandemic. Clin Infect Dis. 2018 Jul 18;67(3):341-349. doi: 10.1093/cid/ciy088. PMID 29746631
- [Derived] Lynfield R, Davey R, Dwyer DE, Losso MH, Wentworth D, Cozzi-Lepri A, Herman-Lamin K, Cholewinska G, David D, Kuetter S, Ternesgen Z, Uyeki TM, Lane HC, Lundgren J, Neaton JD; INSIGHT Influenza Study Group. Outcomes of influenza A(H1N1)pdm09 virus infection: results from two international cohort studies. PLoS One. 2014 Jul 8;9(7):e101785. doi: 10.1371/journal.pone.0101785. eCollection 2014. PMID 25004134
- See also: INSIGHT website — http://www.insight-trials.org